CLINICAL TRIAL: NCT03179540
Title: Phase II Study to Assess the Safety of Non-operative Management for Low Rectal Cancer
Brief Title: Non-operative Management for Locally Advanced Rectal Cancer
Acronym: NOM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PJT - 148730
Record Dates: First submitted 2017-05-12; First posted 2017-06-07 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Rectal Neoplasms
Keywords: Low Rectal Cancer; Complete Clinical Response; Non-operative Management
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- non-operative management (Experimental): Patients with low rectal cancer who have achieved a complete clinical response following chemoradiotherapy will undergo active follow-up with regular clinical visits, physical exam, endoscopy and imaging assessments at regular intervals for 2 years to assess for tumour re-growth or spread to the liver and lungs
  Interventions: Procedure: Non-operative management

INTERVENTIONS:
Procedure: Non-operative management — Patients who are eligible and provide informed consent to participate in the trial will undergo non-operative management (i.e., active surveillance for 24 months) according to the schedule outlined in the study protocol.

SUMMARY:
This is a 5 year Phase II study to evaluate the safety of non-operative management (NOM) in patients with low rectal cancer (LRC) who achieve a complete clinical response (cCR) following chemoradiotherapy (CRT). The safety of NOM will be evaluated by assessing (i) rate of local re-growth and (ii) rate of macroscopically positive resection margin (R2) when surgery is required due to local re-growth. NOM will be considered safe or as effective as surgery to achieve local control if the rate of local re-growth is equal to or less than 30% and the rate of a macroscopically positive margin is 0%.

DETAILED DESCRIPTION:
Background: The standard treatment for low rectal cancer (LRC) involving the anal sphincter involves combined, pre-operative chemotherapy and radiotherapy (CRT) followed by surgery. Surgery involves removal of the rectum and anus and creation of a permanent colostomy and has significant long term effects on bowel and sexual function and body image. Because of the high morbidity of surgery, there has been increasing interest in non-operative management (NOM) for LRC. The NOM approach involves deferral of surgery and active surveillance of all patients with LRC who have achieved a complete clinical response (i.e., have no residual tumour) following completion CRT which occurs in approximately 30% of patients. To date, while there have been a few, prospective single institution studies that have shown favourable results with NOM, this approach has not been adopted into clinical practice due to concerns from physicians about the safety of NOM based on the limited evidence available.

Objectives: Therefore, the objective of this study is to conduct a pan-Canadian Phase II trial to assess the safety of NOM for LRC.

Methods: All patients with LRC requiring surgery and a permanent colostomy being treated at the participating centres will be assessed for complete clinical response (cCR) eight to ten weeks following the completion of CRT by the treating surgeon. For the study, a cCR will be defined as (i) no palpable tumour on digital rectal exam, (ii) no residual tumour defined as white-yellow, flat scar on endoscopy, (iii) no residual tumour on MRI, (iv) no suspicious mesorectal or extramesorectal lymph nodes on MRI and (v) normal CEA level. Patients who meet all of these criteria for cCR will be invited to participate in the study. Patients who consent to participate in the study will undergo active surveillance that will include DRE, endoscopy and pelvic MRI every 3, 6, 9, 12, 18 and 24 months; CEA levels every 3, 6, 9, 12, 15, 18, 21, 24 months and CT chest/abdomen and pelvis every 6, 12, 18 and 24 months. The primary outcome for the study will be the rate of local re-growth 2 years following the completion of CRT. Local re-growth will be defined as failure to meet the cCR criteria at any time point. NOM will be considered safe, if the rate of local re-growth is less than 30% two years after the completion of CRT. The secondary outcomes for the study will be the rate of distant recurrence, disease free and overall survival at 2 years.

Significance: The results of this study will be highly clinically relevant since it is expected that NOM for LRC will be safe and will have significant potential to change clinical practice in Canada and North America since approximately 30% of patients with LRC would be able to safely avoid surgery and a permanent colostomy and have improved bowel and sexual function and body image. Furthermore, widespread adoption of NOM has the potential to increase health care capacity and decrease treatment costs by reducing the number of surgeries, hospital admissions and costs associated with both surgery and long term surgical morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Completed chemoradiotherapy (CRT) as standard of care [Stage II and Stage III (T3-T4N0, AnyTN1-2)]; [50 Gy (2 Gy x 25 fractions) with 5-FU or capecitabine]
* Planned or probable APR
* ALL criteria for complete clinical response are met between 8 and 10 weeks following completion of CRT
* 18 years or older
* Provides written consent

Exclusion Criteria:

* Unable to undergo MRI
* Metastatic disease (including extramesorectal and retroperitoneal lymph nodes)
* Pregnancy
* Inflammatory bowel disease
* More than one primary colorectal cancer
* Other malignancy within 5 years of treatment for current rectal cancer
* Unfit for surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-03-16 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Rate of local re-growth | 2 years
  The safety of non-operative management will be evaluated by assessing the rate of local re-growth in the study population. This approach will be considered safe if the local re-growth rate is equal to or less than 30%.
Rate of macroscopically positive resection margin | 2 years
  The safety of non-operative management will be evaluated by assessing the rate of macroscopically positive resection margin following surgery in the study population. This approach will be considered safe if the rate is 0%.

SECONDARY OUTCOMES:
Rate of overall survival | 2 years
  Rate of overall survival in the study population assessed 2 years after completion of CRT
Rate of disease-free survival | 2 years
  Rate of disease-free survival in the study population assessed 2 years after completion of CRT
Colostomy-free survival | 2 years
  Rate of colostomy-free survival in the study population assessed 2 years after completion of CRT
Quality of Life | 6, 12, 24 months
  Quality of life will be measured using the EORTC C30 questionnaire and will be assessed at 6, 12 and 24 months.
Bowel Function | 6, 12, 24 months
  Bowel function will be measured using the MSKCC Bowel Function Instrument and will be assessed at 6, 12 and 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Kennedy, Principal Investigator — Sinai Health System
Locations (1):
- Sinai Health System, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No